CLINICAL TRIAL: NCT06858527
Title: Adults With Attention Deficit Hyperactivity Disorder / Substance Use Disorder Comorbidity in Integrated Treatment: Effectiveness and Feasibility
Brief Title: Deficit Hyperactivity Disorder / Substance Use Disorder Comorbidity in Integrated Treatment
Acronym: ATTenTIFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APHP240417; 2023-A02246-39 (Other: IDRCB number)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Substance-related Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Substance-Related Disorders; Cognitive Behavioral Therapy; Dual Diagnosis; Randomized Controlled Trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: All participants receive a group psychotherapeutic intervention of Integrated CBT lasting eight weekly two-hour sessions, in parallel with their usual individual care. The sessions are led by a psychologist trained and certified in the practice of CBT and a psychiatrist specialized in addiction medicine. The psychotherapeutic intervention follows a fixed structure and is inspired by the CBT manual for the management of ADHD associated with SUDs published by Matthys et al. (2018). This intervention includes modules on planning and organization, time and distraction management, emotional regulation, work on impulsive behaviors and social skills, cognitive work, as well as substance use management and relapse prevention.
  The sessions will be punctuated by regular breaks to ensure participants' comfort and the integration of the skills worked on during the sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment-Waiting (Other): For this arm, participants receive eight weekly sessions of CBT integrated group treatment in addition to TAU, and then eight weeks of TAU.
  Then, 3 months follow-up, receiving TAU.
  Interventions: Other: TAU+integrated group CBT
- Waiting-Treatment (Other): For this arm, participants receive eight weeks of TAU, and then eight weekly sessions of CBT integrated group treatment in addition to TAU Then, 3 months follow-up, receiving TAU.
  Interventions: Other: TAU+integrated group CBT

INTERVENTIONS:
Other: TAU+integrated group CBT — TAU+integrated group CBT : participants receive a group psychotherapeutic intervention of Integrated CBT lasting eight weekly two-hour sessions, in parallel with their usual individual care. The sessions are led by a psychologist trained and certified in the practice of CBT and a psychiatrist specialized in addiction medicine. The psychotherapeutic intervention follows a fixed structure and is inspired by the CBT manual for the management of ADHD associated with SUDs published by Matthys et al. (2018). This intervention includes modules on planning and organization, time and distraction management, emotional regulation, work on impulsive behaviors and social skills, cognitive work, as well as substance use management and relapse prevention.
  The sessions will be punctuated by regular breaks to ensure participants' comfort and the integration of the skills worked on during the sessions.
  TAU : participants receive their usual care, in exception of group psychotherapeutic interventions.

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) and Substance Use Disorders (SUDs) is a highly common comorbid condition associated with serious medical and psychosocial consequences. However, and despite the international consensus recommending integrated treatment for this comorbidity, few studies tested the efficacy of specific psychotherapeutic treatment for this comorbidity.

The aim of this study is to test the efficacy of a specific group Cognitive and Behavioral Therapy (CBT) for the treatment of adults with this comorbidity.

This is a longitudinal, randomized controlled intervention study utilizing a crossover design between the intervention and treatment-as-usual (TAU) waitlist condition, aimed at testing the effectiveness of an integrated psychotherapeutic group treatment for adults with comorbid Attention Deficit Hyperactivity Disorder (ADHD) and Substance Use Disorders (SUDs).

DETAILED DESCRIPTION:
Substance Use Disorders (SUDs) affect between 0.5% and 15% of the general population and are responsible for a huge morbidity, mortality and social costs (Aldridge et al., 2018; Peterson et al., 2021). Among existing psychotherapeutic approaches, Cognitive and Behavioural Therapy (CBT) is one of the most widely validated, particularly in the addictive population (Hampel et al., 2020; Kabisa et al., 2021; Knapp et al., 2021; Marlatt & Donovan, 2005; Ray et al., 2020). Psychiatric comorbidities are very often associated with SUD (Toftdahl et al., 2016). Among these, Attention Deficit Hyperactivity Disorder (ADHD) is one of the most common, occurring in more than 20% of adults with SUDs (Rohner et al., 2023; van Emmerik-van Oortmerssen et al., 2012) compared with 2.6% in the general population (Song et al., 2021).

The diagnosis and management of adult ADHD are difficult (Cortese et al., 2018; Lopez et al., 2018), particularly when ADHD is comorbid with SUD (Fatséas et al., 2016; Icick et al., 2020; Young et al., 2015). No specific treatment has been yet validated for this comorbidity. It is noteworthy that recognition of adult ADHD has grown considerably in France over the last years.

In this field, the international consensus on the screening, diagnosis and management of this comorbidity recommends integrated treatments (targeting the different disorders at the same time), combining pharmacotherapy with psychotherapy, emphasing the relevance of CBT in this field (Crunelle et al., 2018; Özgen et al., 2020). Despite these immense unmet needs, only one specific ADHD-SUDs psychotherapeutic program has been evaluated to date (van Emmerik-van Oortmerssen et al., 2019)

This protocol aims to test the efficacity of an integrated group Cognitive Behavioral Therapy (CBT) treatment for adults with comorbid Attention Deficit Hyperactivity Disorder (ADHD) and Substance Use Disorders (SUDs) on emotional dysregulation at the primary outcome. Addiction and ADHD symptoms, quality of life, self-esteem, and transdiagnostic constructs (impulsivity, perseverative thinking) are considered as secondary outcomes.

This study corresponds to a longitudinal intervention study using a cross-over design between the group intervention and treatment-as-usual (TAU) waiting condition.

Participants corresponding to inclusion criteria and consenting to participate are enrolled to the study and undergo a first interview assessing clinical and sociodemographic variables and self-rated questionnaires for primary and secondary outcomes. Then they are computer-randomised, controlling for duration of pharmacological treatment in two arms: (1) Treatment-Waiting and (2) Waiting-Treatment. In each condition (Waiting or Treatment) participant conserve their usual treatment for SUD and ADHD, excluding psychotherapeutic group interventions.

The first sequence consists in eight weeks of treatment (TAU for the Waiting-Intervention arm, and TAU+integrated group CBT for the Intervention-Waiting arm). The integrated group CBT consists in weekly two hours groups sessions. At the end of the first sequence and before the second sequence, participants undergo again self-report questionnaires for primary and secondary outcomes.

For the second sequence, participants switch the intervention condition for eight weeks (TAU+integrated group CBT for the Waiting-Intervention arm, and TAU for the Intervention-Waiting arm). At the end of this sequence, participants undergo again self-report questionnaires for primary and secondary outcomes, representing (1) post-intervention data for the Waiting-Intervention arm and (2) a two moths follow-up for the Intervention-Waiting arm.

The third sequence (follow-up) consists in three months of TAU condition, without any exclusion criteria for psychotherapeutic group interventions, ending with a last completion of a shortened battery of questionnaires for primary and secondary outcomes (if needed, questionnaires could be assessed by phone).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older ;
* Suffer from at least one moderate to severe SUD regarding the DSM-5 (tobacco excluded) ;
* Being currently treated for a SUD by a physician of a psychologist ;
* Being diagnosed with an ADHD according to the DIVA 2.0 of DIVA-5 ;
* Being affiliated to a health insurance ;
* Understanding and being able to express himselves in French
* Signed consent

Exclusion Criteria:

* Age under 18;
* Pregnant or breastfeeding women;
* Not having sign the consent form;
* Major difficulties in understanding and/or expressing themselves in french;
* Severe cognitive impairment;
* Acute medical condition making assessment impossible and/or contraindicating participation in group intervention;
* Substance use disorder in a protected environment, currentlu or in the last 15 days, or expected during the study;
* No substance use disorder other than tobacco use disorder;
* Persons under guardianship;
* Participant deprived of liberty or under penal care orders;
* Participation in another group psychotherapeutic intervention throughout the duration of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Emotion dysregulation | Week 1 ; Week 9 ; Week 18 ; Week 31
  Emotion dysregulation subscale of the Adult Self Report Scale for ADHD ( ASRS-31). The scale score ranges from 0 (low dysregulation) to 16 (high dysregulation).

SECONDARY OUTCOMES:
Substance use | Week 1 ; Week 9 ; Week 18 ; Week 31
  Description: Frequency and quantity of substance in the last 15 days, assessed with the Timeline Follow-Back Questionnaire (TLFB)
Self-confidence in abstinence | Week 1 ; Week 9 ; Week 18 ; Week 31
  Description: Self-confidence in the capacity to not use substance in several tempting contexts, assessed with the Brief Situational Confidence Questionnaire (BSCQ). The scale score ranges from 0% (low self-confidence) to 16 (high self-confidence).
Craving | Week 1 ; Week 9 ; Week 18
  Craving frequency and intensity measured with the Craving Experience Questionnaire (CEQ).The frequency scale ranges from 11 (very infrequent) to 110 (always) and the intensity scale ranges from 11 (low) to 110 (extreme).
Nicotine dependence | Week 1 ; Week 9 ; Week 18 ; Week 31
  Nicotine dependence assessed with the Heaviness of Smoking Index (HSI).The total score ranges from 0 (no dependence) to 6 (severe dependence).
ADHD symptoms | Week 1 ; Week 9 ; Week 18
  ADHD symptoms are assessed with the total score of Adult Self Report Scale for ADHD (ASRS-32) and the four subscales (Inattention, Hyperactivity-Impulsivity, emotion dysregulation and executive functions deficit). ). The total score ranges from 0 (low ADHD severity) to 124 (high ADHD severity). The Inattention subscale ranges from 0 (low inattentive symptoms) to 36 (high inattentive symptoms). The Hyperactive-Impulsive subscale ranges from 0 (low hyperactive-impulsive symptoms) to 36 (high hyperactive-impulsive symptoms). The emotion dysregulation subscale ranges from 0 (low dysregulation) to 16 (high dysregulation). The executive function deficit subscale ranges from 0 (low deficit) to 36 (severe deficit).
Impulsivity | Week 1 ; Week 9 ; Week 18
  Impulsivity is measured with the UPPS-P self-report scale. The UPPS-P total score ranges from 20 (low impulsivity) to 80 (high impulsivity).
Perseverative thinking | Week 1 ; Week 9 ; Week 18
  Ruminations are assessed with the Perseverative Thinking Questionnaire (PTQ), a self-report scale. The total score ranges from 0 (no ruminations) to 40 (severe rumination).
Global Quality of life | Week 1 ; Week 9 ; Week 18 ; Week 31
  Global Quality of life is assessed with a visual analogue scale from 0 (very poor quality) to 100 (very good quality)
Physical Quality of life | Week 1 ; Week 9 ; Week 18 ; Week 31
  Physical quality of life is assessed with a visual analogue scale from 0 (very poor quality) to 100 (very good quality)
Psychological Quality of life | Week 1 ; Week 9 ; Week 18 ; Week 31
  Psychological quality of life is assessed with a visual analogue scale from 0 (very poor quality) to 100 (very good quality)
Self Esteem | Week 1 ; Week 9 ; Week 18
  Self-esteem is measured with a single self-report item : the Self Esteem Single Index (SISE)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Therribout, PhD, Principal Investigator — Paris-Nanterre University, UR-4430 CLIPSYD ; Paris-Cité University, UMR-S-1144 INSERM; Fernand-Widal Hospital AP-HP; Romain Icick, MD, PhD, Study Director — Paris-Cité University, UMR-S-1144 INSERM; Fernand-Widal Hospital AP-HP; Lucia Romo, MD, PhD, Study Director — Paris-Nanterre University, UR-4430 CLIPSYD
Locations (1):
- Hôpital Fernand Widal, Assistance-Publique - Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young JT, Carruthers S, Kaye S, Allsop S, Gilsenan J, Degenhardt L, van de Glind G, van den Brink W, Preen D. Comorbid attention deficit hyperactivity disorder and substance use disorder complexity and chronicity in treatment-seeking adults. Drug Alcohol Rev. 2015 Nov;34(6):683-93. doi: 10.1111/dar.12249. Epub 2015 Mar 18. PMID 25790353
- [Background] van Emmerik-van Oortmerssen K, Vedel E, Kramer FJ, Blankers M, Dekker JJM, van den Brink W, Schoevers RA. Integrated cognitive behavioral therapy for ADHD in adult substance use disorder patients: Results of a randomized clinical trial. Drug Alcohol Depend. 2019 Apr 1;197:28-36. doi: 10.1016/j.drugalcdep.2018.12.023. Epub 2019 Feb 5. PMID 30769263
- [Background] van Emmerik-van Oortmerssen K, van de Glind G, van den Brink W, Smit F, Crunelle CL, Swets M, Schoevers RA. Prevalence of attention-deficit hyperactivity disorder in substance use disorder patients: a meta-analysis and meta-regression analysis. Drug Alcohol Depend. 2012 Apr 1;122(1-2):11-9. doi: 10.1016/j.drugalcdep.2011.12.007. Epub 2011 Dec 30. PMID 22209385
- [Background] Toftdahl NG, Nordentoft M, Hjorthoj C. Prevalence of substance use disorders in psychiatric patients: a nationwide Danish population-based study. Soc Psychiatry Psychiatr Epidemiol. 2016 Jan;51(1):129-40. doi: 10.1007/s00127-015-1104-4. Epub 2015 Aug 11. PMID 26260950
- [Background] Song P, Zha M, Yang Q, Zhang Y, Li X, Rudan I; Global Health Epidemiology Reference Group (GHERG). The prevalence of adult attention-deficit hyperactivity disorder: A global systematic review and meta-analysis. J Glob Health. 2021 Feb 11;11:04009. doi: 10.7189/jogh.11.04009. PMID 33692893
- [Background] Rohner H, Gaspar N, Philipsen A, Schulze M. Prevalence of Attention Deficit Hyperactivity Disorder (ADHD) among Substance Use Disorder (SUD) Populations: Meta-Analysis. Int J Environ Res Public Health. 2023 Jan 10;20(2):1275. doi: 10.3390/ijerph20021275. PMID 36674031
- [Background] Ray LA, Meredith LR, Kiluk BD, Walthers J, Carroll KM, Magill M. Combined Pharmacotherapy and Cognitive Behavioral Therapy for Adults With Alcohol or Substance Use Disorders: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jun 1;3(6):e208279. doi: 10.1001/jamanetworkopen.2020.8279. PMID 32558914
- [Background] Peterson C, Li M, Xu L, Mikosz CA, Luo F. Assessment of Annual Cost of Substance Use Disorder in US Hospitals. JAMA Netw Open. 2021 Mar 1;4(3):e210242. doi: 10.1001/jamanetworkopen.2021.0242. PMID 33666661
- [Background] Ozgen H, Spijkerman R, Noack M, Holtmann M, Schellekens ASA, van de Glind G, Banaschewski T, Barta C, Begeman A, Casas M, Crunelle CL, Daigre Blanco C, Dalsgaard S, Demetrovics Z, den Boer J, Dom G, Eapen V, Faraone SV, Franck J, Gonzalez RA, Grau-Lopez L, Groenman AP, Hemphala M, Icick R, Johnson B, Kaess M, Kapitany-Foveny M, Kasinathan JG, Kaye SS, Kiefer F, Konstenius M, Levin FR, Luderer M, Martinotti G, Matthys FIA, Meszaros G, Moggi F, Munasur-Naidoo AP, Post M, Rabinovitz S, Ramos-Quiroga JA, Sala R, Shafi A, Slobodin O, Staal WG, Thomasius R, Truter I, van Kernebeek MW, Velez-Pastrana MC, Vollstadt-Klein S, Vorspan F, Young JT, Yule A, van den Brink W, Hendriks V. International Consensus Statement for the Screening, Diagnosis, and Treatment of Adolescents with Concurrent Attention-Deficit/Hyperactivity Disorder and Substance Use Disorder. Eur Addict Res. 2020;26(4-5):223-232. doi: 10.1159/000508385. Epub 2020 Jul 7. PMID 32634814
- [Background] Lopez PL, Torrente FM, Ciapponi A, Lischinsky AG, Cetkovich-Bakmas M, Rojas JI, Romano M, Manes FF. Cognitive-behavioural interventions for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2018 Mar 23;3(3):CD010840. doi: 10.1002/14651858.CD010840.pub2. PMID 29566425
- [Background] Knapp KS, Brick TR, Bunce SC, Deneke E, Cleveland HH. Daily meaningfulness among patients with opioid use disorder: Examining the role of social experiences during residential treatment and links with post-treatment relapse. Addict Behav. 2021 Aug;119:106914. doi: 10.1016/j.addbeh.2021.106914. Epub 2021 Mar 16. PMID 33857730
- [Background] Kabisa E, Biracyaza E, Habagusenga JD, Umubyeyi A. Determinants and prevalence of relapse among patients with substance use disorders: case of Icyizere Psychotherapeutic Centre. Subst Abuse Treat Prev Policy. 2021 Feb 1;16(1):13. doi: 10.1186/s13011-021-00347-0. PMID 33526066
- [Background] Icick R, Moggi F, Slobodin O, Dom G, Mathys F, van den Brink W, Levin FR, Blankers M, Kaye S, Demetrovics Z, van de Glind G, Velez-Pastrana MC, Schellekens ASA; ICASA-group. Attention Deficit/Hyperactivity Disorder and Global Severity Profiles in Treatment-Seeking Patients with Substance Use Disorders. Eur Addict Res. 2020;26(4-5):201-210. doi: 10.1159/000508546. Epub 2020 Jun 22. PMID 32570249
- [Background] Hampel B, Kusejko K, Kouyos RD, Boni J, Flepp M, Stockle M, Conen A, Beguelin C, Kunzler-Heule P, Nicca D, Schmidt AJ, Nguyen H, Delaloye J, Rougemont M, Bernasconi E, Rauch A, Gunthard HF, Braun DL, Fehr J; Swiss HIV Cohort Study group. Chemsex drugs on the rise: a longitudinal analysis of the Swiss HIV Cohort Study from 2007 to 2017. HIV Med. 2020 Apr;21(4):228-239. doi: 10.1111/hiv.12821. Epub 2019 Dec 18. PMID 31849182
- [Background] Fatseas M, Hurmic H, Serre F, Debrabant R, Daulouede JP, Denis C, Auriacombe M. Addiction severity pattern associated with adult and childhood Attention Deficit Hyperactivity Disorder (ADHD) in patients with addictions. Psychiatry Res. 2016 Dec 30;246:656-662. doi: 10.1016/j.psychres.2016.10.071. Epub 2016 Nov 1. PMID 27842945
- [Background] Crunelle CL, van den Brink W, Moggi F, Konstenius M, Franck J, Levin FR, van de Glind G, Demetrovics Z, Coetzee C, Luderer M, Schellekens A; ICASA consensus group; Matthys F. International Consensus Statement on Screening, Diagnosis and Treatment of Substance Use Disorder Patients with Comorbid Attention Deficit/Hyperactivity Disorder. Eur Addict Res. 2018;24(1):43-51. doi: 10.1159/000487767. Epub 2018 Mar 6. PMID 29510390
- [Background] Cortese S, Adamo N, Del Giovane C, Mohr-Jensen C, Hayes AJ, Carucci S, Atkinson LZ, Tessari L, Banaschewski T, Coghill D, Hollis C, Simonoff E, Zuddas A, Barbui C, Purgato M, Steinhausen HC, Shokraneh F, Xia J, Cipriani A. Comparative efficacy and tolerability of medications for attention-deficit hyperactivity disorder in children, adolescents, and adults: a systematic review and network meta-analysis. Lancet Psychiatry. 2018 Sep;5(9):727-738. doi: 10.1016/S2215-0366(18)30269-4. Epub 2018 Aug 7. PMID 30097390
- [Background] Aldridge RW, Story A, Hwang SW, Nordentoft M, Luchenski SA, Hartwell G, Tweed EJ, Lewer D, Vittal Katikireddi S, Hayward AC. Morbidity and mortality in homeless individuals, prisoners, sex workers, and individuals with substance use disorders in high-income countries: a systematic review and meta-analysis. Lancet. 2018 Jan 20;391(10117):241-250. doi: 10.1016/S0140-6736(17)31869-X. Epub 2017 Nov 12. PMID 29137869
- [Background] Marlatt, G. A., & Donovan, D. M. (Éds.). (2005). Relapse prevention : Maintenance strategies in the treatment of addictive behaviors (2nd ed). Guilford Press.
- [Background] Matthys, F., Bronckaerts, A., & Crunelle, C. L. (2018). Managing ADHD in the presence of substance use disorders. Gompel & Svacina